CLINICAL TRIAL: NCT01422967
Title: Changes of Sleep on the Sensorimotor and Cytokine in Patients With Knee Osteoarthritis
Brief Title: Changes Of Sleep on the Sensoriomotor and Cytokine In Patients With Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Andressa da Silva de Mello, Msc, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 109/2011
Record Dates: First submitted 2011-08-19; First posted 2011-08-25 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Osteoathritis and Sleep
Keywords: Osteoarthritis; Sleep; muscle strength; balance
MeSH Terms: conditions — Osteoarthritis | interventions — Muscle Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Osteoarthritis group (Active Comparator)
  Interventions: Behavioral: Balance and muscle strength
- without osteoarthritis (Active Comparator)
  Interventions: Behavioral: Balance and muscle strength

INTERVENTIONS:
Behavioral: Balance and muscle strength — Balance test: bi and unipodal balance in the place force Muscle strength: bilateral test of knee in dynamometer isokinetic

SUMMARY:
Osteoarthritis (OA) is one of the major health problems and their prevalence has increased in recent decades. It has been shown that OA causes negative effects on sleep and that these changes in sleep see to be correlated with the function and physical performance of patients with OA. However, no study to date has demonstrated the effects of sleep changes in sensorimotor control and systemic inflammatory response in patients with OA. The objective of this study is to assess the influence of sleep changes in sensorimotor control (postural and neuromuscular control) and inflammatory markers (cytokines) in patients with knee OA grade I or II. Participate in this study, 60 male volunteers, aged between 40 and 65. These volunteers will be divided into four groups: Group 1 (n = 15): Osteoarthritis and good quality sleep, Group 2 (n = 15): Osteoarthritis and poor quality sleep, Group 3 (n = 15): Without good and Osteoarthritis quality of sleep, Group 4 (n = 15): Without Osteoarthritis and poor quality of sleep. All volunteers will perform a polysomnography to detect the presence or not of changes in sleep. Further testing on the isokinetic dynamometer to evaluate the acceleration time, maximum isometric torque and isokinetic concentric and eccentric maximum quadriceps muscle strength and a submaximal test to evaluate neuromuscular control. Also there will be a test on the force platform to assess the uni-and bipedal postural control, as well as respond to the WOMAC questionnaire that assesses the quality of life in patients with OA. Blood will be collected for analysis of inflammatory cytokines (TNF-alpha, IL-1alpha, IL-1beta, IL-6, IL-8, IL-12, IL-10, TGF-beta). The significance level is 5% (p ≤ 0.05).

DETAILED DESCRIPTION:
The experimental design of each volunteer (all groups) will be evaluated by a physician before beginning the study and posteriomente will perform a polysomnography. The day after polysomnography voluntary blood will be collected. A week after the volunteer will perform the balance test (force platform) and the test of strength (isokinetic).

ELIGIBILITY:
Inclusion Criteria:

* with and without osteoartrhitis
* no other health problems
* sedentary

Exclusion Criteria:

- other clinical and neurobiological conditions

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
SLEEP PATTERN | only one night of the evaluation
  Sleep pattern assessed using Polissonography overnight in the Sleep Institute.
  In all of the protocol the patient must attend two days in the laboratory, and a night nescessaria for polysomnography, and two periods during the day to the test of balance and strength
Bipodal and Unipodal Balance | only an assessment
  The balance test will assessed by force plate, the test lasts for thirty minutes.
Isokinetic test of knee | only an assessment
  The isokinetc tets will assessed by isokinetc dynamometer - Biodex Multi-Joint System 3. The test lasts for forty minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Stela Mattiello, PhD, Principal Investigator — UFSCar
Locations (1):
- Centro de Estudos em Psicobiologia e Exercicio, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Silva A, Mello MT, Serrao PR, Luz RP, Ruiz F, Bittencourt LR, Tufik S, Mattiello SM. Influence of Obstructive Sleep Apnea in the Functional Aspects of Patients With Osteoarthritis. J Clin Sleep Med. 2018 Feb 15;14(2):265-270. doi: 10.5664/jcsm.6950. PMID 29351822